CLINICAL TRIAL: NCT04896515
Title: Intensive Nutrition Therapy Compared to Usual Care in Critically Ill Adults: A Randomised Pilot Trial - Muscle (a Sub-study of INTENT)
Brief Title: INTENT-Muscle (A Sub-study of INTENT)
Status: Completed | Type: Observational
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: ANZIC-RC/ER003
Record Dates: First submitted 2021-04-15; First posted 2021-05-21 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Critically Ill
Keywords: Critically ill; Critical illness; Muscle; Nutrition; Intensive care unit; Ward; Ultrasound; Adult
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard Nutrition Arm: In INTENT (the parent study) participants will be randomised to the i) Standard Nutrition or ii) Intensive Nutrition arm. A brief description of each is below.
  In ICU:
  1. After enrolment, patients allocated to the standard nutrition therapy (control) group will commence or continue nutrition via an enteral tube to a target rate according to unit protocol including the use of promotility agents and the placement of nasojejunal feeding tubes if required.
  2. Parenteral Nutrition (PN) will only be used if the above methods have been attempted, or an absolute contraindication to enteral nutrition (EN) develops.
  After ICU:
  1. Nutrition management will be as per usual site management at that hospital.
- Intensive Nutrition Arm: In ICU:
  1. Supplemental PN will be commenced within 2 hours of randomisation. The starting dose will be determined by the amount of energy received in the 24 hours prior to randomisation
  2. The need for the intervention will be based on the adequacy of nutrition provision and assessed daily until ICU discharge
  3. If there is an interruption of EN for greater than 2 hours the PN must be run at 20 kcal/kg calculated body weight until EN is recommenced. After the interruption, EN should be recommenced as per local protocol.
  After ICU:
  1. An intensive nutrition intervention will be provided on the ward.
  The goal of nutrition care across the hospital stay will be to ensure 80-100% of participant's estimated energy requirements are met.
  Interventions: Dietary Supplement: Supplemental parenteral nutrition

INTERVENTIONS:
Dietary Supplement: Supplemental parenteral nutrition — Supplemental parenteral nutrition OLIMEL N12E (Baxter Healthcare Corporation)
  Groups: Intensive Nutrition Arm

SUMMARY:
The currently recruiting randomised controlled trial "Intensive Nutrition Therapy Compared to Usual Care in Critically Ill Adults" (INTENT, NCT03292237) is the first multi-centre trial to compare an intensive, individualised nutrition intervention to standard care for the duration of hospital admission in critically ill patients. INTENT-Muscle, is an observational longitudinal study nested within INTENT. The aim of INTENT-Muscle is to compare longitudinal changes in muscle health (assessed by bioimpedance and muscle ultrasound) in critically ill patients randomised to each arm of INTENT.

DETAILED DESCRIPTION:
Background: Critically ill patients may experience debilitating loss of muscle mass and strength, leading to substantial functional impairments both during and long after hospitalisation. Little is known about what therapies may attenuate deterioration of muscle health (muscle mass and muscle quality) in this setting but nutrition is thought to be important, based on the physiological response to critical illness.

The currently recruiting randomised controlled trial (RCT) "Intensive Nutrition Therapy Compared to Usual Care in Critically Ill Adults" (ClinicalTrials.gov Identifier: NCT03292237) is the first multi-centre trial to provide an individualised nutrition intervention for the duration of hospital admission in critically ill patients. Combining the most promising and novel bedside techniques for objectively measuring muscle health (bioimpedance technology and ultrasound) with a whole hospital nutrition intervention has never been done before, and will provide crucial data to understand the relationship between nutrition delivery and changes in muscularity from ICU admission to hospital discharge.

Aim: To explore changes in muscle health in response to an individualised nutrition intervention and in association with clinical and functional outcomes, using clinically applicable bedside techniques.

Secondary aims:

In both arms of INTENT to:

1. Compare longitudinal changes in bioimpedance variables (fat-free mass, normally hydrated lean tissue, extracellular/intracellular ratio, and variables from Cole modelling) to hospital discharge (or day 28)
2. Compare longitudinal changes in ultrasound variables (mid-upper arm and quadriceps muscle thickness, rectus femoris cross-sectional area, and rectus femoris echogenicity) to hospital discharge (or day 28)
3. Compare clinical and functional outcomes in patients identified as having low muscularity (assessed by ultrasound) at ICU admission
4. Investigate the relationship between bioimpedance and ultrasound variables with clinical and functional outcomes at baseline and over the hospital admission (collected as part of INTENT)

Hypothesis: In critically ill patients receiving individualised nutrition care for the duration of hospital admission (censored at study day 28), declines in phase angle and muscle health will be attenuated compared to patients receiving standard nutritional care.

ELIGIBILITY:
Inclusion Criteria:

* Randomised to the INTENT trial at a participating sub-study site

Exclusion Criteria:

* Patients will be excluded from the sub-study if they have any of the following:

  * A pacemaker or electronic implantable device
  * Missing limb(s)
  * Unable to get adequate separation in the limbs (e.g. severe obesity)
  * Inaccessible site(s) for electrode placement (e.g. major burns, trauma)
  * Broken skin at the site(s) of electrode placement
  * The treating clinician does not believe the study to be in the best interest of the patient
  * Person responsible/Medical treatment decision maker is of non-English speaking background (therefore cannot provide informed consent) Note Before: If the Person responsible/medical treatment decision maker is of English speaking background but the patient is not (and the Person responsible/Medical treatment decision maker speaks the same language as the patient) you may continue assessing the patient for eligibility to INTENT-Muscle as the Person Responsible/Medical treatment decision maker can translate the Patient Information and Consent Form (PICF) and consent discussion with the patient in order to obtain continuing consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixty to eighty critically ill patients from up to 6 participating INTENT sites in Australia and New Zealand will be recruited to INTENT-Muscle
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Phase angle | Hospital admission (censored at study day 28)
  To compare longitudinal changes in phase angle during hospital admission in patients randomised to both arms of INTENT.

SECONDARY OUTCOMES:
Change in bioelectrical impedance spectroscopy (BIS) derived phase angle | Every 7 days during hospital admission (censored to study day 28)
  Change in BIS-derived phase angle from baseline to hospital discharge and every 7 days between
Change in BIS-derived impedance ratio | Every 7 days during hospital admission (censored to study day 28)
  Change in BIS-derived impedance ratio from baseline to hospital discharge and every 7 days between.
Change in BIS-derived fat-free mass | Every 7 days during hospital admission (censored to study day 28)
  Change in BIS-derived fat-free mass (kg) from baseline to hospital discharge and every 7 days between.
Change in BIS-derived normally-hydrated lean tissue | Every 7 days during hospital admission (censored to study day 28)
  Change in BIS-derived normally-hydrated lean tissue (kg) (generated using the Chamney model) from baseline to hospital discharge and every 7 days between.
Change in BIS-derived Cole model variable R infinity to R0 | Every 7 days during hospital admission (censored to study day 28)
  Change in BIS-derived Cole model variable R infinity to R0 from baseline to hospital discharge and every 7 days between.
Change in BIS-derived characteristic frequency (ωc, a Cole model variable) | Every 7 days during hospital admission (censored to study day 28)
  Change in BIS-derived Cole model variable characteristic frequency (ωc) from baseline to hospital discharge and every 7 days between.
Change in BIS-derived membrane capacitance (a Cole model variable) | Every 7 days during hospital admission (censored to study day 28)
  Change in BIS-derived Cole model variable membrane capacitance from baseline to hospital discharge and every 7 days between.
Change in BIS-derived extra-cellular water | Every 7 days during hospital admission (censored to study day 28)
  Change in BIS-derived extracellular water from baseline to hospital discharge and every 7 days between.
Change in BIS-derived intracellular water | Every 7 days during hospital admission (censored to study day 28)
  Change in BIS-derived intracellular water from baseline to hospital discharge and every 7 days between.
Change in ultrasound-derived Rectus femoris cross-sectional area | Every 7 days during hospital admission (censored to study day 28)
  Change in ultrasound-derived Rectus femoris cross-sectional area (cm2) from baseline to hospital discharge and at measurement points (every 7 days during hospital admission).
Change in ultrasound-derived mid-upper arm muscle thickness | Every 7 days during hospital admission (censored to study day 28)
  Change in ultrasound-derived muscle thickness (in centimetres) at the mid-upper arm from baseline to hospital discharge and at measurement points (every 7 days during hospital admission).
Change in ultrasound-derived bilateral quadriceps muscle thickness | Every 7 days during hospital admission (censored to study day 28)
  Change in ultrasound-derived bilateral quadriceps muscle thickness (in centimetres) from baseline to hospital discharge and at measurement points (every 7 days during hospital admission).
Change in ultrasound-derived Rectus femoris echogenicity | Every 7 days during hospital admission (censored to study day 28)
  Change in ultrasound-derived Rectus femoris echogenicity from baseline to hospital discharge and at measurement points (every 7 days during hospital admission).
Muscle mass at ICU admission | Baseline (Enrolment)
  An estimate of whole-body muscularity at ICU admission (enrolment) will be assessed by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Emma J Ridley, PhD, Principal Investigator — Australian and New Zealand Intensive Care Research Centre
Locations (6):
- Australia (5):
  - Blacktown Hospital, Blacktown, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Ballarat Base Hospital, Ballarat, Victoria
  - Frankston Hospital, Frankston, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Auckland Hospital (CVICU), Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided